CLINICAL TRIAL: NCT03576625
Title: Effect of Buglossoides Oil on Recent Chronic Non-injurious Hip and Knee Pain
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Réseau de Santé Vitalité Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HC-NNHPD-230190
Record Dates: First submitted 2018-06-11; First posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2017-09

CONDITIONS: Hip Pain Chronic; Knee Pain Chronic
Keywords: Buglossoides arvensis; vegetable oil; omega-3 fatty acids; participants

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High oleic sunflower oil (HOSO) (Placebo Comparator): 30 ml HOSO emulsion (equivalent to 9.9 ml oil) in a single dose, 56 days
  Interventions: Dietary Supplement: High Oleic Sunflower Oil
- Buglossoides oil emulsion (Experimental): 30 ml Buglossoides oil emulsion (equivalent to 9.9 ml oil) in a single dose, 56 days
  Interventions: Dietary Supplement: Buglossoides Oil

INTERVENTIONS:
Dietary Supplement: High Oleic Sunflower Oil — Consume oil smoothie (emulsified HOSO) with a meal once daily for 9 weeks
  Other Names: HOSO
  Arms: High oleic sunflower oil (HOSO)
Dietary Supplement: Buglossoides Oil — Consume oil smoothie (emulsified Buglossoides oil) with a meal once daily for 9 weeks
  Other Names: Ahiflower
  Arms: Buglossoides oil emulsion

SUMMARY:
The effect of Buglossoides oil emulsion on the intensity of recent chronic knee and hip pain, on plasma and mononuclear blood cells fatty acid profiles and on whole blood Eicosapentaenoic acid production will be investigated.

DETAILED DESCRIPTION:
This study will document the impact of an emulsion of Buglossoides oil on the intensity of recent chronic knee and hip pain. Secondly, the impact of consuming Buglossoides oil on plasma and leukocyte fatty acid profiles will be investigated, thus providing clinical evidence on the efficacy of an emulsion of Buglossoides oil in increasing EPA content. Lastly, a comprehensive analysis of whole blood eicosanoid production following supplementation will provide data on the potential for Buglossoides oil to modulate immune function.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant women, using an effective form of birth control (such as oral contraceptives, injectable contraceptives or the barrier method such as a intrauterine device (IUD) with a spermicide, a diaphragm with a spermicide, a condom with a spermicide or a sponge with a spermicide) for at least 3 months prior to entry into the study and continuing during participation in the study.
2. 18 to 65 years of age, inclusive.
3. Body mass index (BMI) 18 - 39.9 kg/m2
4. Subject has recent (less than 6 months) current chronic (having lasted more than two weeks) knee (one or both) and/or hip pain that is not the result of an acute injury. Pain intensity is 20 mm or higher using a Visual Analog Scale ranging from 0-100 mm.
5. Subject has no planned knee or hip surgery.
6. Subject is willing to avoid alcohol consumption for 24h prior to every clinic visit.
7. The subject will not modify smoking habits during supplementation period.
8. No significant medical conditions that in the opinion of the qualified physician, would preclude the subject's participation in the study.
9. Signed informed consent.
10. Willing to follow all study procedures including study visits, fasting blood draws, stable body weight, normal eating habits, current activity level, and compliance with study preparation.
11. Willing to not consume fish, crustaceans and shellfish for the duration of the study.
12. Willing to avoid taking anti-inflammatory medications (analgesics and NSAIDs) for 24 hours prior to Visits 2 and 5.

Exclusion Criteria:

1. Pregnancy or lactation. Women trying to conceive. Women who will try to conceive who are unwilling to commit to the use of a medically approved form of contraception throughout the study period. Method of contraception must be recorded in the case report file.
2. Has had a diagnosis of rheumatoid arthritis.
3. Individual has a condition the study physician believes would interfere with the participant's ability to provide informed consent, comply with his responsibilities during the study, which might confound the interpretation of the study results or put the person at undue risk.
4. Self-reported medical conditions including an active peptic ulcer, inflammatory bowel disease, or gastrointestinal bleeding and any medical condition or prior gastrointestinal surgery that could influence absorption, metabolism or excretion of the study supplement.
5. History or presence of significant, renal, hepatic, gastrointestinal, pulmonary, biliary, neurological or endocrine disorders.
6. History or presence of cancer in the past 2 yrs, except for non-melanoma skin cancers (e.g. basal or squamous cell carcinoma of the skin).
7. Clinically significant abnormal laboratory test results including but not limited to LDL-cholesterol ≥ 4.1mM, triglyceride levels ≥3.95mM, fasting creatinine ≥ 1.5 mg/dL, ALT or AST ≥ 1.5X the upper limit of normal.
8. Currently being treated for angina, arrhythmia and/or congestive heart failure. History of myocardial infarction or stroke.
9. Uncontrolled hypertension (resting systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
10. Type 1 or 2 diabetes. Fasting glucose ≥ 100 mg/dL. HbA1c ≥ 6.0.
11. If a smoker, subject smokes no more than 1 pack (20 cigarettes) daily.
12. History (within 12 months) or current alcohol or substance abuse (no more than 14 consumptions per week; 1 consumption= 12 oz beer, 5 oz wine, 1.5 oz distilled spirits).
13. Use of steroidal anti-inflammatory medications (prednisone, etc)
14. Use of any lipid-altering medications (statins, bile acid sequestrants, cholesterol absorption inhibitors, fibrates, prescription formulations of niacin).
15. Unstable use of thyroid medication. Stable, treated hypothyroidism is not an exclusion criteria.
16. Use of any weight loss or lipid metabolism medication/supplement/program (including lipase inhibitors) within 1 month of study period OR weight gain or loss > 2 kg in the past 3 months.
17. Currently taking fish oil or any other omega-3 or omega-6 PUFA supplement/drug within one month of Visit 1 and throughout the study. Consumption of fatty fish (salmon, herring, mackerel, albacore tuna, and sardines) more than 2X a month within one month of visit 1 and throughout the study period. Consumption (more than twice a month) of any EPA/DHA enriched foods (e.g. DHA-enriched eggs) within one month of Visit 1. Unwillingness to avoid all fish including shellfish and crustaceans throughout the study period.
18. Use of alpha-linolenic acid-containing seeds and oils such as flax seed, chia seed, perilla seed, hemp, spirulina, walnut, mustard seed or black currant seeds/oil within one month of Visit 1 and throughout the study.
19. Use of an investigational product within the previous 30 days.
20. Has donated blood up to 4 weeks before the start of the study. Not willing to cease being a blood donor during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in the nature of pain severity | Baseline, 19, 38, 56 days
  Defined by visual analogue scale (VAS)
Change in the nature of fatigue severity | Baseline, 19, 38, 56 days
  Defined by visual analogue scale (VAS)

SECONDARY OUTCOMES:
Nature and frequency of analgesic use | 56 days
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain, stiffness and physical function scores | Baseline, 19, 38, 56 days
Plasma eicosapentaenoic concentration (EPA) | Baseline and day 56
  Expressed as umol/L plasma
Plasma 20:4n-3 | Baseline and day 56
  Expressed as umol/L plasma
Plasma docosapentaenoic acid | Baseline and day 56
  Expressed as umol/L plasma
Plasma 20:4n-3, EPA and DPA individually as % of total fatty acids | Baseline and day 56
Mononuclear cell 20:4n-3, EPA and DPA individually as % of total fatty acids | Baseline and day 56
Eicosanoid profile following ex vivo whole blood immune challenge | Baseline and day 56

CONTACTS AND LOCATIONS:
Overall Officials: Marc Surette, PhD, Principal Investigator — Université de Moncton, Moncton, NB, Canada
Locations (1):
- Université de Moncton, Moncton, New Brunswick, Canada